CLINICAL TRIAL: NCT04229875
Title: Effects of Specialized Treatment for Bipolar Disorder - the CAG Bipolar RCT
Brief Title: The CAG Bipolar the CAG Bipolar RCT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mental Health Centre Copenhagen, Bispebjerg and Frederiksberg Hospital (Other)
Collaborators: Maria Faurholt-Jepsen, MD, DMSc (Unknown); The Mental Health Services in the Capital Region of Denmark (Unknown)
Responsible Party: Principal Investigator, Lars Vedel Kessing, Prof., Principal Investigator, Mental Health Centre Copenhagen, Bispebjerg and Frederiksberg Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H-19067248
Record Dates: First submitted 2020-01-03; First posted 2020-01-18 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: Bipolar Disorder
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CAG Bipolar (Experimental): 1. Patients will be treated in a localized CAG Bipolar clinic within each psychiatric centre increasing the number of bipolar patients for each clinician
  2. All clinicians will get certified in diagnosing and treating bipolar disorder by joining an educational course and ongoing courses continuously
  3. Treatment will include a group-based psychoeducation program
  4. Coordinated targets to improve quality of life of patients by increasing concordance between clinicians, patients and relatives on well-defined treatment goals
  5. Continued ongoing supervision of patient cases in CAG Bipolar staff by the Copenhagen Affective Disorder Clinic
  6. Three-month bidirectional exchange of two clinical staff members between the Copenhagen Affective Disorder Clinic and each CAG Bipolar clinic
  7. Recovery mentors
  Interventions: Other: CAG Bipolar
- Control group (No Intervention): Standard treatment

INTERVENTIONS:
Other: CAG Bipolar — See description of CAG Bipolar
  Arms: CAG Bipolar

SUMMARY:
The CAG Bipolar study is a large-scale pragmatic randomized controlled trial aiming to investigate whether specialized and more centralized treatment (into a clinical academic group (CAG)) improves lives and outcomes for patients with bipolar disorder (N= 1000 patients).

DETAILED DESCRIPTION:
Bipolar disorder is a complex illness with a complex treatment that differs during manic, depressed and remitted states, frequently leaving patients with decreased quality of life and impaired psychosocial function. Traditionally, psychiatry has been sparsely subspecialized in Denmark as well as internationally during the last four decades leaving patients in generalized psychiatric settings. At the same time, demands to clinical skills, research and education have increased, and IT solutions have emerged as a possible way to optimize treatment.

Effects of organizational changes and digital health interventions are rarely investigated scientifically in health care services. This is a randomized controlled trial conducted in the entire Mental Health Services, Capital Region of Denmark including all psychiatric centers in the region.

The CAG Bipolar study is a large-scale pragmatic randomized controlled trial aiming to investigate whether specialized and more centralized treatment (into a clinical academic group (CAG)) improves lives and outcomes for patients with bipolar disorder (N= 1000 patients). Findings from the study will have great impact on future organization and optimization of treatment within psychiatry in Denmark as well as internationally.

ELIGIBILITY:
Inclusion Criteria:

* All patients with a main diagnosis of bipolar disorder in the five largest psychiatric centers in the Mental Health Services, Capital Region of Denmark (Psychiatric Center Copenhagen, Psychiatric Center Hillerød, Psychiatric Center Amager, Psychiatric Center Glostrup and Psychiatric Center Ballerup) will be asked for participation

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2020-01-13 (Actual); Primary Completion 2023-11-13 (Estimated); Study Completion 2025-01-13 (Estimated)

PRIMARY OUTCOMES:
Risk of psychiatric hospitalization | During the entire study period of 12 months pr participant
  Data on hospitalization according to data from the population-based Danish Psychiatric Central Research Register will be collected and analyzed with survival statistics. Assessed blinded for the intervention status
Cumulated duration of hospitalization according to data from the population-based Danish Psychiatric Central Research Register | During the entire study period of 12 months pr participant
  Data on cumulated duration of hospitalization according to data from the population-based Danish Psychiatric Central Research Register will be collected and analyzed with survival statistics. Assessed blinded for the intervention status

SECONDARY OUTCOMES:
Quality of life according to WHO Quality of Life-BREF (WHOQoL) | Baseline, 6 months and 12 months
  Scored between 0-100. Higher scores indicate higher quality of life. Patient evaluated
Perceived stress according to Cohen's Perceived stress scale | Baseline, 6 months and 12 months
  Patient evaluated. Scores between 0-40. Higher score indicate higher perceived stress.
Satisfaction with care according to scores on the Verona Satisfaction Scale-Affective Disorder | Baseline, 6 months and 12 months
  Patient evaluated. Higher scores indicate higher satisfaction with treatment.
Satisfaction with care according to scores on the Danish nation-wide patient satisfaction questionnaire | Baseline, 6 months and 12 months
  Patient evaluated. Higher scores indicate higher satisfaction with treatment.
Adherence to the Danish national guidelines of medical treatment of bipolar disorder according to use of the three main maintenance mood stabilizers for bipolar disorder: lithium, lamotrigine or quetiapine | During the entire study period of 12 months per participant
  Data collected from electronic patient records.
Clinicians' satisfaction with their work at start and end of the RCT | Baseline and 12 months
  Clinician evaluated using the Medical Personnel Job Satisfaction Questionnaire
Patient-reported depressive symptoms according to the major depressive Inventory (MDI) | Baseline, 6 months and 12 months
  Patient-evaluated. Higher scores indicate higher level of depressive symptoms.
Patient-reported manic symptoms according to the Altman Self-rating Scale for Mania (ASRM) | Baseline, 6 months and 12 months
  Patient-evaluated. Higher scores indicate higher level of manic symptoms.
Proportion of patients starting group-based psychoeducation | During the entire study period of 12 months per centre
  Proportion of patients in clinics starting in group-based psychoeducation

OTHER OUTCOMES:
Long-term register-based outcome measures: risk of hospitalization | 3, 5 and 10 years follow-up
  Danish registry data with data available on number of longt-term hospitalizations
Long-term register-based outcome measures: duration of hospitalization | 3, 5 and 10 years follow-up
  Danish registry data with data available on number of longt-term days during hospitalizations
Long-term register-based outcome measures: prescribed medication | 3, 5 and 10 years follow-up
  Danish registry data with data available on the medicine prescribed
Long-term register-based outcome measures: psychosocial measures (sickdays) | 3, 5 and 10 years follow-up
  Danish registry data with data available on number of days away form work
Long-term register-based outcome measures: somatic comorbidity | 3, 5 and 10 years follow-up
  Danish registry data with data available on somatic diagnoses
Long-term register-based outcome measures: rate of suicide and death | 3, 5 and 10 years follow-up
  Danish registry data with the data available

CONTACTS AND LOCATIONS:
Locations (1):
- Psychiatric Center Copenhagen, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kessing LV, Kyster NB, Bondo-Kozuch P, Christensen EM, Vejstrup B, Smidt B, Jorgensen AB, Rosenberg R, Mardosas D, Rasmussen LB, Vinberg M, Hageman I, Faurholt-Jepsen M; CAG Bipolar Study group. Effect of specialised versus generalised outpatient treatment for bipolar disorder: the CAG Bipolar trial - study protocol for a randomised controlled trial. BMJ Open. 2021 Oct 13;11(10):e048821. doi: 10.1136/bmjopen-2021-048821. PMID 34645661